CLINICAL TRIAL: NCT06782061
Title: A Pilot Study on the Activation of NOD2 Receptors in Preterm Infants by Lactobacillus Reuteri DSM17938
Brief Title: Activation of NOD2 Receptors in Preterm Infants by Lactobacillus Reuteri DSM17938
Acronym: NOD2-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NFEC-2024-654
Record Dates: First submitted 2024-12-24; First posted 2025-01-17 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Preterm Infants
Keywords: DSM17938; NOD2; preterm infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Parallel
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DSM17938+Routine clinical treatment (Experimental): Lactobacillus reuteri DSM17938，5 drops per day by mouth (containing at least 100 million CFU of Lactobacillus reuteri DSM17938)
  Interventions: Other: DSM17938+Routine clinical treatment
- Routine clinical treatment (No Intervention): Routine clinical treatment

INTERVENTIONS:
Other: DSM17938+Routine clinical treatment — Lactobacillus reuteri DSM17938，5 drops per day by mouth (containing at least 100 million CFU of Lactobacillus reuteri DSM17938)，Routine clinical treatment
  Arms: DSM17938+Routine clinical treatment

SUMMARY:
Primary Objective: To evaluate the capacity of Lactobacillus reuteri DSM17938 to activate NOD2 receptors in preterm infants.

Secondary Objective: To analyze the impact of Lactobacillus reuteri DSM17938 on the gut microbiome of preterm infants

DETAILED DESCRIPTION:
This study was designed as an open-label, stratified, randomized, parallel-controlled pilot study, using gestational age as the stratification factor. Participants were stratified according to birth gestational age < 32 weeks, 32 weeks ≤ birth gestational age < 37 weeks, and simple randomization method was used in each gestational age group. All subjects were enrolled after birth/hospital admission, and the experimental group started intervention at 10-14 days after birth, and the intervention period was 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants with a gestational age of less than 37 weeks.
2. Birth weight of less than 2500 grams.
3. Hospitalized within 72 hours after birth.
4. Parents or legal guardians have signed an informed consent form.

Exclusion Criteria:

1. Congenital digestive tract malformations, genetic metabolic diseases, or congenital immunodeficiency diseases.
2. A history of severe asphyxia, infection, or liver and kidney dysfunction at birth/enrollment.
3. Death within 72 hours after birth.

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2024-12-26 (Actual); Primary Completion 2025-01-19 (Actual); Study Completion 2025-01-19 (Actual)

PRIMARY OUTCOMES:
Concentration of NOD2 ligand in fecal samples | Pre-intervention Phase: On the 3rd day after birth (V1), 7th day (V2), and 10th day (V3). Intervention Phase: During the intervention period, on the 2nd day (V4), 4th day (V5), 6th day (V6), 8th day (V7), 10th day (V8), 12th day (V9), and 14th day (V10)
  The supernatants of fecal samples were used to examine the content of NOD2 ligand with the human NOD2/NF-κB/secreted embryonic alkaline phosphatase (SEAP) reporter HEK293 cell

SECONDARY OUTCOMES:
Relative Abundance of Operational Taxonomic Units (OTUs) in Fecal Samples | Pre-intervention Phase: On the 3rd day after birth (V1), 7th day (V2), and 10th day (V3). Intervention Phase: During the intervention period, on the 2nd day (V4), 4th day (V5), 6th day (V6), 8th day (V7), 10th day (V8), 12th day (V9), and 14th day (V10)
  DNA extraction was performed using the QIAamp Mini Kit following the manufacturer's instructions. The V4 hypervariable region of the 16S ribosomal RNA (rRNA) gene was amplified and sequenced on an Illumina ISEQ 100 platform, generating 250 bp paired-end reads. Raw sequencing data quality was assessed and controlled using fastp (v0.23.2). Adapter sequences corresponding to the V3-V4 region were removed with cutadapt. Amplicon sequence variants (ASVs) were identified by denoising the paired-end FASTQ files with DADA2 (v1.6.0) in R. Representative sequences were aligned using the PyNAST algorithm (v1.2.2), and a phylogenetic tree was constructed with FastTree (v2.1.3). Taxonomic classification of ASVs was performed using the Ribosomal Database Project (RDP) classifier against the Greengenes database. To minimize biases from variations in sequencing depth, all samples were rarefied before downstream analyses.
Concentration of DSM17938 per Gram of Feces Quantified by qPCR | Pre-intervention Phase: On the 3rd day after birth (V1), 7th day (V2), and 10th day (V3). Intervention Phase: During the intervention period, on the 2nd day (V4), 4th day (V5), 6th day (V6), 8th day (V7), 10th day (V8), 12th day (V9), and 14th day (V10)
  Quantitative fluorescence PCR (qPCR) was used to detect DSM17938

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shen, Doctor, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The following study documentation will be made available for sharing: study protocol, statistical analysis plan, informed consent form, clinical study report, and analytic code.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The study data will be accessible for sharing during a specified temporal window, initiating three months after study completion and publication, with availability extending through a two-year period post-publication.
Access Criteria: Data can be shared with researchers for scientific purposes upon application to the corresponding author. The research institution's ethics committee and data safety committee will review such requests. Data sharing will be permitted only following committee approval and after proper de-identification of patient information.
URL: https://www.ncbi.nlm.nih.gov/